CLINICAL TRIAL: NCT03677193
Title: Biofeedback-enhanced Interactive Computer-play for Youth With Cerebral Palsy: a Feasibility Pilot Study Measuring the Effect of Play on Wrist and Hand Activity
Brief Title: Biofeedback-enhanced Interactive Computer-play for Youth With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-785
Record Dates: First submitted 2018-07-31; First posted 2018-09-19 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: The study will be conducted a single-case experimental design (SCED). Participants will be randomly assigned to begin the intervention at staggered starting-points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental)
  Interventions: Behavioral: Playing ICP game

INTERVENTIONS:
Behavioral: Playing ICP game — Participants will play the ICP game from their home this is expected to be 30 min * 5 days / week for 4 weeks. Once per week, participants will play the ICP game with a researcher.

SUMMARY:
The protocol aims to evaluate the feasibility and potential efficacy of an Interactive Computer Play (ICP) intervention. The ICP intervention is built to help youth with Cerebral palsy (CP) who have difficulty performing activities of daily living with their hand.

The ICP intervention is a video game controlled by performing gestures with the non-dominant hand. Using Low-cost commercial technology muscle activity and arm movement is used to recognize the gestures which control the game. Players will get feedback in the game about the quality of their movements through the built-in points and rewards system. This repetitive practice and feedback will help the participants build strength and control in their arm. To evaluate this ICP intervention, 10 participants, with hemiplegic CP and 8-18 years old, from Holland Bloorview will be recruited for a pilot feasibility study using a single-case experimental design (SCED). The design is as follows:

1. Phase 1. Participants will speak with therapists / researchers in an Initial Dialogue to:

   1. Introduce the study/game and what it offers types of daily activities
   2. Set Performance goal areas (Canadian Occupational Performance Measure (COPM)), and
   3. Develop an action plan to facilitate the successful achievement of their goals.
2. Phase 2. Participants will perform baseline functional assessments including: active range of motion (AROM), Assisting Hand Assessment (AHA), Box and Blocks Test (B&B).
3. Phase 3. During the 4-week intervention, participants will play the ICP game from their home according to the goals they define during the initial dialogue. This is expected to be 20-30 min * 5 days per week. Once per week, participants will play the ICP intervention with a researcher in clinic or at home who will also measure AROM while recording the play session.
4. Phase 4. After the intervention, participants will complete clinical measures of functional performance (AROM, AHA, B&B) a final time and speak with therapist and researcher to re-evaluate goals (COPM).

By leveraging the motivational and immersive aspects of ICP and combining it with evidence-based movement feedback this protocol has the potential to improve home-based ICP therapies for persons with CP.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of Cerebral Palsy.
2. Age: 8-18 years. This age range was selected given the popularity of video games and the size of the muscle sensors available.
3. Manual Abilities Classification System levels I-III.
4. Have a goal relating to improving hand / wrist function.
5. Dominantly spastic presentation
6. Able to co-operate, understand, and follow simple instructions for game play. This will be assessed during the information and assent process by the researcher.
7. Having passive ROM of at least 10° greater than AROM.

Exclusion Criteria:

1. History of unmanaged epilepsy. Video game systems are not recommended for individuals with a history of epilepsy as per manufacturer's Health and Safety Precautions.
2. Has received a Botulinum Toxin treatment within 3 months or constraint-based movement therapy within 6 months of the study enrollment.
3. Visual, cognitive or auditory disability at a level that would interfere with game play. The child must have normal or corrected to normal vision and hearing.
4. Dominantly dystonic presentation
5. Unable to commit an estimated minimum of 10 hours to their training plan over four weeks.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-03-14 (Actual); Study Completion 2019-03-15 (Actual)

PRIMARY OUTCOMES:
Change in Active Range of Motion (AROM) | pre-intervention, each week of intervention (weeks 1-4 of the intervention)
  active wrist AROM
Change in Canadian Occupational Performance Measure (COPM) | pre-intervention, post-intervention (5 weeks after pre-intervention)
  Evaluates changes in perceived function and satisfaction of performance in self-identified goal areas.

SECONDARY OUTCOMES:
Change in Assisting Hand Assessment (AHA) | Pre-intervention, post-intervention (5 weeks after pre-intervention)
  a sequence of bimanual tasks through the semi-structured progression of a board game (~15 minutes).
Change in Box and Blocks Test (B&B) | Pre-intervention, post-intervention (5 weeks after pre-intervention)
  the participant has one minute to move blocks from one side of a box, over a center divider, and place on the other side of the box.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Biddiss, PhD, Principal Investigator — Bloorview Research Institute
Locations (1):
- Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] MacIntosh A, Desailly E, Vignais N, Vigneron V, Biddiss E. A biofeedback-enhanced therapeutic exercise video game intervention for young people with cerebral palsy: A randomized single-case experimental design feasibility study. PLoS One. 2020 Jun 22;15(6):e0234767. doi: 10.1371/journal.pone.0234767. eCollection 2020. PMID 32569284